CLINICAL TRIAL: NCT02388048
Title: A Phase II Study of the Combination of Ofatumumab and Ibrutinib Followed by Allogeneic Bone Marrow Transplant or Consolidation for Pretreated High Risk Patients With Chronic Lymphocytic Leukemia
Brief Title: Ofatumumab & Ibrutinib + Allogeneic Bone Marrow Transplant or Consolidation in High Risk Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LLC1215; 2015-000684-13 (EudraCT Number)
Record Dates: First submitted 2015-03-09; First posted 2015-03-13 (Estimated); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Leukemia, Lymphoblastic, Chronic
Keywords: Leukemia; Chronic; High-risk; ofatumumab; ibrutinib; Lymphoblastic
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia; Bronchiolitis Obliterans Syndrome | interventions — ibrutinib; ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ibrutinib + Ofatumumab (Experimental): IBRUTINIB 420 mg PO daily in 28-day cycles for a total of 7 cycles (28 weeks).
  OFATUMUMAB 300 mg on day 1 of cycle 2 of Ibrutinib, followed by 2000 mg on D8, 15, 22 of cycle 2, D1, 8, 15, 22 of cycle 3, and Day 1 of cycle 4-7.
  After induction treatment patients with HLA identical sibling or fully matched MUD donor will be addressed to reduced intensity allogeneic bone marrow transplant, while patients without a suitable donor or who refuse the transplant procedure will receive maintenance treatment by BTK inhibitor (IBRUTINIB 420 mg PO daily in 28-day cycles). Treatment will continue until disease progression or unacceptable toxicity.
  Interventions: Drug: Ibrutinib + ofatumumab

INTERVENTIONS:
Drug: Ibrutinib + ofatumumab

SUMMARY:
A clinical study to evaluate a treatment with two drugs, named Ofatumumab and Ibrutinib, in patients with lymphoblastic acute leukemia who have been already treated with other therapies.

DETAILED DESCRIPTION:
This is a phase II multicenter, non-comparative, open label study for high risk previously treated patients with CLL, requiring therapy, aimed at evaluating the efficacy of the Ofatumumab and Ibrutinib combination.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18 years or until 65 years;
2. Confirmation of B-CLL previously treated with no more than 1 previous line of treatment .
3. Risk patients with CLL defined as follows:

   * treated patients showing 17p deletion in >20% of the cells by FISH, or TP53 mutation or,
   * resistant (SD/PD) to fludarabine containing combination therapy or relapse within 12 months from a fludarabine-containing combination therapy.
4. Active disease meeting at least 1 of the following IWCLL criteria for requiring treatment:

   * Evidence of progressive marrow failure as manifested by the development of, or worsening of anemia (Hb< 10 g/dL) and/or thrombocytopenia (platelets < 100,000/mL).
   * Massive (≥ 6 cm below the left costal margin), progressive, or symptomatic splenomegaly.
   * Massive nodes (at least 10 cm longest diameter), or progressive or symptomatic lymphadenopathy.
   * Progressive lymphocytosis with an increase of more than 50% over a 2-month period or a lymphocyte doubling time (LDT) of < 6 months.
   * Autoimmune hemolytic anemia and/or immune thrombocytopenia that is poorly responsive to corticosteroids or other standard therapy.
   * One or more disease-related symptoms:
   * unintentional weight loss > 10% within 6 months prior to screening;
   * significant fatigue (inability to work or perform usual activities);
   * fevers >38.0°C for 2 or more weeks prior to screening;
   * night sweats for more than 1 month prior to screening.
5. Stage B or C of CLL according to Binet staging system;
6. Stage A disease fitting the criteria for treatment according to the IWCLL-NCI criteria (2008) are also included.
7. WHO performance status 0-II.
8. Life expectancy ≥ 6 months.
9. Hematology values must be within the following limits:

   * Absolute neutrophil count (ANC) ≥ 750/mm3 independent of growth factor support;
   * Platelets ≥100,000/mm3 or ≥ 30.000/mm3 if bone marrow involvement independent of transfusion support in either situation.
10. Biochemical values within the following limits:

    * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x upper limit of normal (ULN).
    * Total bilirubin ≤ 1.5 x ULN unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin.
    * Serum creatinine ≤ 2 x ULN or estimated Glomerular Filtration Rate (Cockroft Gault) ≥ 30 mL/min/1.73m2.
11. Women of childbearing potential and men who are sexually active must be practicing a highly effective method of birth control during and after the study For females, these restrictions apply for 1 month after the last dose of ibrutinib and for 12 months after the last dose of Ofatumumab. For males, these restrictions apply for 3 months after the last dose of ibrutinib. Men must agree to not donate sperm during and after the study.
12. Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [β-hCG]) or urine pregnancy test at Screening. Women who are pregnant or breastfeeding are ineligible for this study.
13. Sign an informed consent document indicating that they understand the purpose of and procedures required for the study, including biomarkers, and are willing to participate in the study.

Exclusion Criteria:

1. Major surgery within 3 weeks before registration.
2. Known central nervous system lymphoma.
3. History of stroke or intracranial hemorrhage within 6 months prior to registration.
4. Requires anticoagulation with warfarin or equivalent vitamin K antagonists (eg, phenprocoumon).
5. Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification.
6. Vaccinated with live, attenuated vaccines within 4 weeks of registration.
7. Known history of human immunodeficiency virus (HIV) or active Hepatitis C Virus or active Hepatitis B Virus infection or any uncontrolled active systemic infection requiring intravenous (IV) antibiotics.
8. Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of ibrutinib capsules, or put the study outcomes at undue risk.
9. Positive serology for Hepatitis B (HB) defined as a positive test for HBsAg. In addition, if negative for HBsAg but HBcAb positive (regardless of HBsAb status), a HBDNA test will be performed and if positive the subject will be excluded. ***see attached monitoring criteria for HBcAb+ and HBV DNA negative subjects.
10. Other past or current malignancy. Subjects who have been free of malignancy for at least 5 years, or have a history of completely resected non-melanoma skin cancer, or successfully treated in situ carcinoma are eligible.
11. Requirement for treatment with a strong CYP3A4/5 and/or CYP2D6 inhibitor.
12. Significant concurrent, uncontrolled medical condition including, but not limited to, renal, hepatic, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease which in the opinion of the investigator may represent a risk for the patient.
13. Inability to swallow capsules or tablets, or disease significantly affecting gastrointestinal function and/or inhibiting small intestine absorption.
14. Chronic or current infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment such as, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis, tuberculosis.
15. Uncontrolled autoimmune hemolytic anemia or idiopathic thrombocytopenic purpura.
16. Central nervous system involvement with CLL.
17. Subjects who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment).
18. Treatment with any known non-marketed drug substance or experimental therapy within 5 terminal half lives or 4 weeks prior to enrollment, whichever is longer, or currently participating in any other interventional clinical study.
19. Prior treatment with anti-CD20 monoclonal antibody or alemtuzumab within 3 months prior to the start of therapy.
20. History of significant cerebrovascular disease in the past 6 months or ongoing event with active symptoms or sequelae.

    * If HBV DNA is negative, subject may be included but must undergo at least every 2 month HBV DNA PCR testing from the start of treatment during the treatment course. Prophylactic antiviral therapy may be initiated at the discretion of the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-10; Primary Completion 2024-04-03 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
The number of pretreated patients with high risk CLL who achieve a Complete Response (CR) after the induction therapy with Ibrutinib plus Ofatumumab. | After 6.5 years from treatment start

SECONDARY OUTCOMES:
Number of patients in Complete Response (CR)/Partial Response (PR) | After 28 weeks from treatment start
  Overall response rate at the end of induction therapy.
Number of patients without progression of the disease. | At 60 months from treatment start
  Progression-free survival
Number of patients alive | At 60 months from treatment start
  Overall survival
Number of patients without events | At 60 months from treatment start
  Event-free survival
Number of Minimal Residual Disease-negative Complete Responses | At 28 weeks from treatment start
  6. To estimate Minimal Residual Disease (MRD) in terms of rate of MRD-negative CRs at the end of induction therapy and after SCT or Ibrutinib maintenance therapy for patients in CR
Number of adverse events | At 6.5 years after treatment start
  7. Safety profile and tolerability of the combination of Ofatumumab and Ibrutinib and the ibrutinib as maintenance in terms of type, frequency, severity and relationship of adverse events (AEs).

CONTACTS AND LOCATIONS:
Overall Officials: Marco Montillo, Study Chair — Department of Hematology, Niguarda Ca' Granda, Milan; Francesca R. Mauro, Study Director — Department of Hematology, Policlinico Umberto I di Roma
Locations (35):
- Italy (35):
  - Università degli Studi "Sapienza" - Dip Biotecnologie Cellulari ed Ematologia - Divisione di Ematologia, Roma, Provincia
  - S.O.C. di Ematologia - Azienda Ospedaliera - SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - Area Vasta N. 5 Ascoli Piceno - S. Benedetto Del Tronto, Presidio Ospedaliero Av5 Osp. Gen. Prov.Le "C.G.Mazzoni" - Uoc Ematologia, Ascoli Piceno
  - Nuovo Record Esporta in Excel Stampa Esporta in file di testo Mostra Informazioni Record Multi edit Stato dello studio presso il centro records: 28 Record 1/28 su 28 direzione di ordinamento Centro (CIC) direzione di ordinamento Sperimentatore Pri, Bologna
  - ASL N.8 - Ospedale "A. Businco" - Struttura Complessa di Ematologia e CTMO, Cagliari
  - Università di Catania - Cattedra di Ematologia - Ospedale "Ferrarotto", Catania
  - Azienda Ospedaliera Pugliese Ciaccio - Presidio Ospedaliero A.Pugliese - Unità Operativa di Ematologia, Catanzaro
  - Nuovo Record Esporta in Excel Stampa Esporta in file di testo Mostra Informazioni Record Multi edit Stato dello studio presso il centro records: 28 Record 1/28 su 28 direzione di ordinamento Centro (CIC) direzione di ordinamento Sperimentatore Pri, Cona
  - U.O. Ematologia - P.O. Annunziata - A.O. di Cosenza, Cosenza
  - Policlinico di Careggi, Florence
  - IRCCS_AOU San Martino-IST-Ematologia 1-Monoblocco 11°piano- lato ponente, Genova
  - ASL Le/1 P.O. Vito Fazzi - U.O. di Ematologia ed UTIE, Lecce
  - Istituto Scientifico Romagnoli per lo Studio e la Cura dei Tumori- IRST, Meldola
  - Divisione di Ematologia - Azienda Ospedaliera Ospedali Riuniti "Papardo Piemonte" P.O. Papardo, Messina
  - Aulss 3 Serenissima, Ospedale Dell'Angelo - Mestre - Uo Ematologia, Mestre
  - Fondazione Irccs "Istituto Nazionale Tumori" - Milano - Sc Ematologia, Milan
  - Ospedale Niguarda " Ca Granda" - SC Ematologia Blocco SUD, Ponti Est, Scala E, 4° piano, Milan
  - S.C.D.U. Ematologia - DIMECS e Dipartimento Oncologico - Università del Piemonte Orientale Amedeo Avogadro, Novara
  - Aou Di Padova - Uo Ematologia, Padua
  - Sl Salerno, Presidio Ospedaliero Tortora Pagani - Ematologia, Pagani
  - U.O. di Ematologia con trapianto - Centro di Riferimento Regionale per le coagulopatie rare nel bambino e nell'adulto Dipart. Biomedico di Medicina Interna - A.U. Policlinico "Paolo Giaccone", Palermo
  - Cattedra di Ematologia CTMO Università degli Studi di Parma, Parma
  - Sezione di Ematologia ed Immunologia Clinica - Ospedale S.Maria della Misericordia, Perugia
  - U.O. Ematologia Clinica - Azienda USL di Pescara, Pescara
  - Asl Di Piacenza, Ospedale "Guglielmo Da Saliceto" - Ematologia E Centro Trapianti, Piacenza
  - Unità Operativa Complessa di Ematologia - Arcispedale S. Maria Nuova, Reggio Emilia
  - Ospedale "Infermi", Rimini
  - Università Cattolica del Sacro Cuore - Policlinico A. Gemelli, Roma
  - Università degli Studi - Policlinico di Tor Vergata, Roma
  - Università Degli Studi Di Roma "Sapienza" - Dipartimento Di Medicina Traslazionale E Di Precisione - U.O.C. Ematologia, Roma
  - A.O. Santa Maria - Terni S.C Oncoematologia, Terni
  - A.O. Mauriziano Umberto I, Torino
  - Dipartimento di Oncologia ed Ematologia S.C. Ematologia 2 A.O. Città della Salute e della Scienza di Torino San Giovanni Battista, Torino
  - Divisione di Ematologia dell' Università degli Studi di Torino - "Città della Salute e della Scienza di Torino", Torino
  - Università degli Studi di Verona - A. O. - Istituti Ospitalieri di Verona- Div. di Ematologia - Policlinico G.B. Rossi, Verona

IPD SHARING:
Plan to Share IPD: No